CLINICAL TRIAL: NCT06113939
Title: A Randomized Controlled Pilot Trial Comparing 2 Non-invasive Airway Clearance Methods for the Prevention of Early-onset Ventilator-associated Pneumonia.
Brief Title: Prevention of Infection of the Respiratory Tract Through Application of Non-Invasive Methods of Secretion Suctioning
Acronym: PIRAMIDES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Miguel Sanchez Garcia, Director Critical Care Department, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PIRAMIDES
Record Dates: First submitted 2023-10-10; First posted 2023-11-02 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Intubation Complication; Stroke, Ischemic; Stroke Hemorrhagic; Head Trauma; Cardiac Arrest; Ventilator Associated Pneumonia; Airway Clearance Impairment
Keywords: ventilator-associated pneumonia; prevention; airway clearance
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Craniocerebral Trauma; Heart Arrest; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: Open label randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of Care (Active Comparator): IV ceftriaxone/24 hours 3 doses
  Interventions: Device: airway clearance
- Subglottic aspiration (Experimental): Continuos aspiration of subglottic secretions
  Interventions: Device: airway clearance
- Cough Simulator (Experimental): Mechanical exsufflator
  Interventions: Device: airway clearance

INTERVENTIONS:
Device: airway clearance — mechanical suctioning of airway secretions

SUMMARY:
Severe trauma, head trauma, stroke and resuscitated cardiac arrest patients requiring endotracheal intubation and mechanical ventilation are at high risk of early-onset ventilator-associated pneumonia (EO-VAP). A short course of systemic antibiotic is recommended for prophylaxis.

This study intends to assess the safety and efficacy of 2 alternative mechanical non-invasive airway clearance techniques in the prevention of EO-VAP in an open label randomized pilot trial of 20 subjects per study group i.e., 60 cases. The interventions will be in place for 7 days and the observational periods will be 14 days.

DETAILED DESCRIPTION:
Background. Patients with structural coma are at high risk of so-called early onset pneumonia (EOP). Incidence rates of up to 50% have been reported in patients with head trauma or stroke. The usual causative microorganisms belong to the normal upper airway flora like Streptococcus pneumoniae, Staphylococcus aureus, Haemophilus influenza and Moraxella catarrhalis. EOP typically is not present at admission and develops after 2 to 7 days after endotracheal intubation.

A short course of systemic antibiotic therapy and aspiration of subglottic secretions (ASS) are associated with significant reductions in EOP, although ASS does not prevent late-onset pneumonia. Non-invasive mechanical methods may avoid the use of prophylactic antibiotics and pain and injury to the tracheal mucosa caused by the conventional suctioning catheter.

The primary objectives of the present randomized pilot trial is to compare the prevention of respiratory tract infections during invasive mechanical ventilation and occurrence of device-associated adverse events of non-invasive mechanical airway clearance devices with standard of care in the ICU Department at Hospital Clinico San Carlos.

Secondary objectives are duration of intubation and respiratory support (mechanical intubation plus high flow nasal cannula).

Methods. Informed consent will be requested from relatives in patients admitted to intensive care (Neuro-trauma unit) requiring endotracheal intubation estimated to last >48 hours, who do not have a hopeless prognosis.

Closed envelopes will be used for allocation to one of the 3 study groups::

1. Control group: ceftriaxone 2 g/24 hours, 3 doses
2. Subglottic aspiration of secretions
3. Cough simulator

Patients in all groups will receive the topical components of selective decontamination of the digestive tract (SDD) while intubated.

In groups 2 and 3 the allocated study group prevention intervention will be applied during the first 7 days.

The main study objectives will be monitored over the first 14 days of intubation or until extubation if performed before day 14.

Sample size will be 60 subjects, 20 per study group, enrolled in blocs of 5, with the 5th case of each bloc being allocated in random sequence.

Nurses will be trained in using the devices for groups 2 and 3 before the start of enrollment phase.

The diagnosis of pneumonia vs tracheobronchitis will be based on chest x-ray and confirmed by lung ultrasound to exclude chest x-ray false negatives.

On day 5 to 7 or immediately before extubation, if planned earlier, electrical impedance tomography will be performed to compare lung air distribution and compliance between groups.

ELIGIBILITY:
Inclusion Criteria:

* Endotracheal intubation anticipated to last >48 hours
* Stroke
* Severe Trauma
* Head Trauma
* Resuscitated cardiac arrest

Exclusion Criteria:

* Ominous prognosis
* Limitation of Life support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-19 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Incidence density of Respiratory tract infection per 1000 days of intubation | inclusion to day 14
  ventilator-associated pneumonia or tracheobronchitis
Incidence of adverse events | inclusion to day 14
  Device-related complications

SECONDARY OUTCOMES:
Duration of Respiratory support | inclusion until ICU discharge or death
  Duration of mechanical ventilation plus high-flow nasal cannula
Systemic antibiotic use | inclusion to day 14
  Number of patients needing antibiotic therapy for respiratory tract infection and antimicrobial DDDs
Incidence and type of Bacterial resistance | 14 days
  Identification of resistance bacteria in respiratory tract samples

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Alvarez-Gonzalez, MD.PhD, Study Director — Hospial Clinico San Carlos; Sandra Garcia Pintado, RN, Principal Investigator — Hospial Clinico San Carlos
Locations (1):
- Hospital Clinico San Carlos, Madrid, Madrid, Spain